CLINICAL TRIAL: NCT03886376
Title: Effects of Systematic Massage Application on Swimming Athletes Performance: a Randomized, Placebo-controlled Clinical Trial
Brief Title: Systematic Massage on Swimming Athletes Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Flávia Carvalho, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018/09680-8
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Athletes
Keywords: Athletes; Swimming; Performance; Massage

STUDY DESIGN:
Intervention Model Description: For the control group, immediately after the resistance training the athletes were instructed to wait for 12 minutes until the beginning of the swimming training. The deep massage group received 12 minutes of massage on the legs, arms and the back with three different sliding pressures. The superficial massage group received superficial massage on the same sites than the intervention group. The three conditions were performed after a resistance training and before a swimming training.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Massage (Experimental): The deep massage was performed three times during a training week, after a physical training and before the swimming training
  Interventions: Other: Deep Massage
- Superficial Massage (Active Comparator): The superficial massage was performed three times during a training week, after a physical training and before the swimming training
  Interventions: Other: Superficial Massage
- Control (No Intervention): The control group kept their normal routine of training. Immediately after the physical training the athletes were instructed to wait for 12 minutes (passive recovery) until the beginning of the swim training.

INTERVENTIONS:
Other: Deep Massage — The deep massage group received 12 minutes of massage on the legs, arms and the back with three different sliding pressures.
  Arms: Deep Massage
Other: Superficial Massage — The superficial massage group received 12 minutes of only one sliding pressure performed on the legs, arms and the back.
  Arms: Superficial Massage

SUMMARY:
Swimming is a sport that includes different styles and distances, which can expose the athlete to different stressors that can affect performance and generate conditions such as overtraining. This is due to the lack of integration of systematic recovery periods during training programs. A very used recuperative feature in swimming is massage. Recent studies have shown that the application of short duration is sufficient to obtain the desired effects and it is possible that its application systematized over a period of time may have greater effects on performance. The aims of this study were to evaluate the effects of deep and superficial massage on clinical, functional and performance issues; to identify its short-term effects on clinical and functional variables and to investigate the association between training load and the swimmer's perceptions.

DETAILED DESCRIPTION:
The study was composed by a convenience sample of 19 male and female athletes aged between 12 and 20 years old who train regularly (six days a week) and are members of the Prudentina Athletic Sports Association (APEA) swimming team. The research project was accepted by the Research Ethics Committee of the Faculty of Science and Technology of the Paulista State University "Júlio de Mesquita Filho" - FCT / UNESP. A single-blinded crossover randomized controlled trial with 1:1:1 allocation. The sample was submitted to a balanced-block randomization, by sorting on Excel, with a balanced sex, age and competitive level ratio, to three sequences of interventions containing: (i) control, (ii) superficial massage and iii) deep massage. The study was conducted over a period of eight weeks, consisting of five sessions of resistance and swimming training. The option for intervention time point was based on a pilot study that yielded higher training loads on on Mondays, Tuesdays and Fridays and worse perceptions between both training stimuli (resistance and swimming). At the end of each training week, participants were subjected to a maximum test of 100-m front crawl sprint in a semi-olympic indoor pool (25 meters), then we performed a functional evaluation. Training load was monitored over the entire trial by the Session Rating of Perceived Exertion (sRPE) calculated by the product of the training duration and perception of effort. Effects of single massage on perceptive outcomes were analyzed by generalized estimating equations (GEE) with ordinal distribution and cumulative logit link function, using intervention group, training time-points and day of intervention as predictors in the model. The first category (nothing) was used as reference unless otherwise stated. Effects of repeated massage on proprioception was analyzed by GEE and remaining outcomes were analyzed by Generalized Linear Mixed Model, both with Gamma distribution and cumulative logit link function. Bonferroni adjustments were used for all significant main effect. Pearson's test was used to explore the correlation between training load and performance and interpreted as small (0.00-0.25), fair (0.26-0.50), moderate to good (0.51-0.75) and excellent (>0.75).

ELIGIBILITY:
Inclusion Criteria:

* regular members of the Prudentina Association of Athletic Sports (APEA)
* between 12 and 20 years old

Exclusion Criteria:

* not attending the evaluation session

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Adjusted Performance | up to 1 week
  Technical index (FINA points)
Performance | up to 1 week
  Sprint time (s)

SECONDARY OUTCOMES:
Inferior limb power | up to 1 week
  Squat jump test (cm)
Superior limb power | up to 1 week
  Bench press test (m/s)
Flexibility | up to 1 week
  Tested by hip flexion measured by the centimeters reached on the Wells bench
Proprioception | up to 1 week
  Laser-pointer assisted angle reproduction test for 55°, 90° and 125° of shoulder flexion
Perceptions | up to 1 week
  Swimmer's Perception of Effort Questionnaire (SPEQ) composed of 5 perceptions (well-being, heaviness, tiredness, discomfort, pain) rated by a 1-5 likert scale where 1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely. For well-being higher values indicate better outcomes while for the remaining perceptions higher values indicate worse outcomes
Swimming velocity | up to 1 week
  Swimming velocity (SV) is derived from the central 10m of the pool and the time to swim this distance (t), calculated by the formula SV=10/t.
Stroke frequency | up to 1 week
  Stroke frequency (SF) is derived from the number os strokes (n) and the time to swim the central 10m of the pool (t), calculated by the formula SF=n/t.
Distance per stroke | up to 1 week
  Distance per stroke (DPS) is derived from the swimming velocity and swimming frequency, calculated by the formula DPS=SV/SF.
Stroke index | up to 1 week
  Stroke index (SI) is derived from the swimming velocity and the distance per stroke, calculate from the formula SI=SV*DPS.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Pastre, doctor, Study Director — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Sao Paulo State University, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared because they belong to a competitive team and most of the participants have less than 18 years old